CLINICAL TRIAL: NCT03456193
Title: Allogeneic Left Atrial and Pulmonary Vein Transplant for Pulmonary Vein Stenosis
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: reviewing eligibility criteria
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, David Hoganson, Instructor in Cardiac surgery, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00023581
Record Dates: First submitted 2018-02-22; First posted 2018-03-07 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Pulmonary Vein Stenosis
MeSH Terms: conditions — Stenosis, Pulmonary Vein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LA transplantation (Experimental): The left atrium and pulmonary veins will be transplanted into the recipient
  Interventions: Procedure: LA transplant

INTERVENTIONS:
Procedure: LA transplant — The proposed study treatment will include three central components:
  * Harvest of the left atrium and pulmonary veins from a suitable donor
  * Excision of the left atrium and portions of stenotic pulmonary veins from the patient with pulmonary vein stenosis
  * Implantation of the donor posterior left atrium and portions of pulmonary veins into the patient.

SUMMARY:
This is a prospective, single center, safety and feasibility trial to evaluate the transplantation of the left atrium and pulmonary veins in patients with pulmonary vein stenosis. Consented patients will be listed for transplantation. Once a suitable donor has been identified, the left atrium, pulmonary veins and complete lung block will be harvested from the donor and transported to Boston Children's Hospital as is the procedure for routine lung transplantation patients. The left atrium and pulmonary veins will be transplanted into the recipient. The recipient will receive the normal immunosuppression protocol used for heart transplantation.

This pilot study will include 5 patients.

DETAILED DESCRIPTION:
Techniques for harvest of the posterior left atrium and pulmonary veins from a suitable organ donor have been well established as this is currently accomplished during every harvest of lungs for lung transplantation. The difference in this therapy is that the lung parenchyma will not be utilized. However, the harvest from the donor will be exactly the same with the full lung block typically harvested for lung transplant removed and transported back to the site of implantation. The exact extent of pulmonary vein utilization from the lung block will be determined at the time of implantation based on the exact anatomy and location of the pulmonary vein disease of the recipient.

As this represents a new transplantation approach, this program has been discussed with the United Network for Organ Sharing (UNOS) and the New England Organ Bank (NEOB). UNOS identified this as a new area of transplantation related to but separate from heart or lung transplantations. Eventually if this progresses to a national phase, it will require creation of a new patient waiting list and all the policies that accompany a new area of transplantation. Although there is enthusiasm at UNOS for this approach, they recommended that it be pursued as a regional research program as an initial step. The NEOB also has voiced support for this program in a meeting with them including their medical director. They are interested in supporting this program as a Region 1 research program and will perform a full evaluation for approval once local IRB approval has been granted. The Children's team will work closely with NEOB to create a list of potential patients and identify suitable donors.

Utilizing standardized harvesting techniques will minimize any changes to the current harvest approach and definition of tissue allocation during the harvest procedure. As the lung parenchyma is unnecessary, it is expected that suitable donors for left atrial transplant would come from two sources:

* The first source is brain dead donors in whom the lungs are not allocated for transplantation based on rejection of the lungs for quality or no matching donors.
* The second source is donors after cardiac death (DCD) which are utilized in the adult population for kidney, liver and lung transplantation. DCD organs are not currently utilized pediatric lung transplantation. However, as the viability of these tissues, including the entire lung block is well established, these represent a potential donor pool for left atrial transplant patients.

Certainly experience with preservation of the kidney grafts for hours or days with integrated perfusion systems has demonstrated the successful implantation of vascularized tissues appropriately preserved can be extended beyond the traditional four hour window targeted for lung transplantation. Kidney transplants are commonly done within 24 hours without evidence of impact on the vascular patency these grafts. In addition, only vascular tissue is being transplanted that has no effect on gas exchange or contractility. Accordingly it is expected that the goal implantation time for left atrial transplants after harvest will not need to be within the four to six hour window used for lung transplant but can be safely extended to 24 hours. This window extends the donor pool for left atrial transplants to the entire country.

Excision of recipient left atrium and stenotic pulmonary veins and implantation of left atrial graft The set up for the operation will be identical to all major cardiopulmonary bypass cardiac cases. The surgical approach for the recipient will likely be a clamshell incision that crosses the sternum in the fourth interspace. This is the same incision used for lung transplant. The patient will be cannulated for cardiopulmonary bypass in the distal aorta, SVC and low in the IVC. Cardiopulmonary bypass will be initiated and the patient will be cooled to 18°C. Prior to arresting the heart, the donor left atrium and pulmonary veins will be inspected in the lung block. The pulmonary veins from the donor will be mobilized and prepared for resection from the lung block.

The cross clamp will be applied and the heart arrested. The pulmonary veins of the recipient will be mobilized and transected beyond the level stenoses. The left atrium and pulmonary vein graft then be brought to the field and positioned in the orthotopic position.

The anastomosis of the pulmonary veins will be completed with a generous diameter of the anastomotic area to minimize any risk of late anastomotic narrowing even in the smallest of pulmonary vein segments. The donor left atrium will be anastomosed to the posterior left atrial cuff of the heart. Only the affected pulmonary veins with stenosis will be transplanted. This may be one or up to all 4 main pulmonary veins. If an individual pulmonary vein or side of pulmonary veins are unaffected, they will not have any manipulation or intervention on them. A formal atrial fenestration will be created. Post-bypass evaluation with transesophageal echocardiogram will assess pulmonary vein velocities and flow. The chest will be closed and patient transferred intubated to the ICU.

In the initial clinical experience with these transplants, a traditional immunosuppression protocol for heart transplants will be followed. Over time new protocols will be developed and tested which focused on minimizing the long-term immunosuppression regimens.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary vein stenosis involving at least one but up to all of the main pulmonary veins following initial treatment, including but not limited to balloon dilation, stenting, surgical repair or chemotherapy
* Focal pulmonary stenosis limited to the main pulmonary veins or their first or second order branches.

Exclusion Criteria:

* Diffuse pulmonary vein stenosis involving long segments of one or more pulmonary veins including diffuse stenosis into the second order pulmonary vein branches or beyond
* Significant underlying lung disease
* Irreversible pulmonary artery hypertension exceeding indexed 10 Woods units (WU)
* Irreversible multisystem organ failure; or additive effects of multiple systems affected making transplant survival unlikely
* Progressive systemic disease with early mortality (genetic/metabolic, idiopathic, syndromic)
* Morbid obesity (BMI>30)
* Diabetes mellitus with evidence of end-organ damage
* Severe chromosomal, neurologic or syndromic abnormalities
* Active infection
* HIV or chronic hepatitis B or C infection
* Severe left ventricular dysfunction
* Malignancy within 5 years prior to transplant
* Severe renal or liver failure
* Inadequate social support for post-transplant management
* Recent history of illicit drug, tobacco or alcohol abuse despite trials/assistance to stop behavior
* Episode of acute rejection within the previous 6 months
* Post-transplant lymphoproliferative disease that has been within two years
* Evidence of large stroke with high risk for hemorrhagic conversion

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Short term survival | 30 days
  Mortality rate at 30 days following transplantation.

SECONDARY OUTCOMES:
Pulmonary vein patency | 30 days
  The study team will assess for the flow through the transplanted pulmonary veins.
Long term survival | 6 months
  Mortality rate at 6 months following transplantation.
Long term pulmonary vein patency and gradient | 6 months
  The study team will assess for the flow through the transplanted pulmonary veins and any increased gradient through the transplanted pulmonary veins (gradient through transplanted veins that has been deemed greater than mild).
Right ventricular pressure | 6 months
  The study team will assess for any increase in right ventricular pressure and/or concerns for developing pulmonary hypertension.

CONTACTS AND LOCATIONS:
Overall Officials: David Hoganson, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Devaney EJ, Chang AC, Ohye RG, Bove EL. Management of congenital and acquired pulmonary vein stenosis. Ann Thorac Surg. 2006 Mar;81(3):992-5; discussion 995-6. doi: 10.1016/j.athoracsur.2005.08.020. PMID 16488708
- [Background] Yun TJ, Coles JG, Konstantinov IE, Al-Radi OO, Wald RM, Guerra V, de Oliveira NC, Van Arsdell GS, Williams WG, Smallhorn J, Caldarone CA. Conventional and sutureless techniques for management of the pulmonary veins: Evolution of indications from postrepair pulmonary vein stenosis to primary pulmonary vein anomalies. J Thorac Cardiovasc Surg. 2005 Jan;129(1):167-74. doi: 10.1016/j.jtcvs.2004.08.043. PMID 15632839
- [Background] Bharat A, Epstein DJ, Grady M, Faro A, Michelson P, Sweet SC, Huddleston CB. Lung transplant is a viable treatment option for patients with congenital and acquired pulmonary vein stenosis. J Heart Lung Transplant. 2013 Jun;32(6):621-5. doi: 10.1016/j.healun.2013.03.002. PMID 23701851
- [Background] Sadr IM, Tan PE, Kieran MW, Jenkins KJ. Mechanism of pulmonary vein stenosis in infants with normally connected veins. Am J Cardiol. 2000 Sep 1;86(5):577-9, A10. doi: 10.1016/s0002-9149(00)01022-5. PMID 11009286